CLINICAL TRIAL: NCT01904591
Title: The Effects of Anti-oxidants on Clinical Outcomes and Radiological Features of Chronic Spinal Cord Injury: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Paul Stacey, Clinical Scholar/ Fellow: Physical Medicine and Rehabilitation, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCIantiox1
Record Dates: First submitted 2013-07-10; First posted 2013-07-22 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Antioxidants; tractography; ASIA assessment
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Selenium; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selenium and Vitamin E (Experimental): single arm, all subjects receive both vitamins for 1 year from time zero.
  Interventions: Dietary Supplement: Selenium; Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Selenium — Selenium 50 micrograms daily per oral
  1 year of treatment
  Other Names: brand to be determined.
Dietary Supplement: Vitamin E — Vitamin E 400 international units daily per oral
  1 year of treatment
  Other Names: Brand to be determined

SUMMARY:
This study will enroll 10 adults with a chronic spinal cord injury. The investigators will image their damaged motor tracts using MRI tractography scanning, and the investigators will formally assess their ASIA motor level at the outset of the study. Then, the investigators will treat them with one year of 'over the counter' dosage of selenium and vitamin E. These are two vitamins known to be anti-oxidants. After one year the investigators will repeat the MRI scans and ASIA assessments to determine if their has been any change in the appearance of motor tracts on MRI tractography, or in motor level on ASIA exam. As this is a pilot study the investigators are primarily concerned with establishing safety of this intervention, with a view to conducting a larger and more rigorous controlled trial in the future. The investigators also have a small hope that in fact some improvement might be found with vitamin treatment.

DETAILED DESCRIPTION:
This is an open label prospective pilot study. The results of this study will assist the researchers in organizing a larger study. The objective of the study is to determine if treatment with over the counter nutrients (Vitamin E and Selenium) may improve recovery in patients with remote traumatic spinal cord injury (SCI). The investigators will enroll 10 adults with remote traumatic spinal cord injury. The participant will have experienced their injury at least one year prior to enrollment, are currently living in the community. Participants may not have any other neurological cause of weakness (i.e. stroke or traumatic brain injury), must be able to undergo MRI scanning, and be able to take the oral medications as prescribed. At the beginning of the study, baseline strength will be measured by a standardized (American Spinal Injury Association) exam. This exam will be repeated one year after taking the treatment. Furthermore specialized radiological imaging (MRI tractography) of the spinal cord will be completed prior to taking the medications, and one year subsequently. MRI tractography is advanced imaging technology that is able to generate quantitive images of the nerve fiber tracts in the spinal cord that control limb movement. We anticipate that treatment with Vitamin E and selenium for a one period year will increase the ASIA motor score and/or increase the nerve density of the nerve tracts in the spinal cord that control limb movement

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Spinal cord injury at least on year prior to enrollment
* Able to swallow pills at described dose and by mouth
* Able to provide informed consent
* Able to travel to Hamilton General Hospital for initial and follow-up MRI tractography studies
* Willing to attend monthly meetings with investigators

Exclusion Criteria:

* Contraindication to MRI scanning such as metal in the body, pacemaker, implanted nerve stimulator, or claustrophobia.
* Concomitant neurological condition such as stroke, acquired brain injury, peripheral nerve injury
* Pressure ulcer at time of enrollment into study
* Uncontrolled autonomic dysreflexia
* Current usage of anticoagulants
* Allergy to Selenium or Vitamin E, or present supplementation of both/ either nutrient at study dosage levels.
* History of Cardiovascular disease (heart attack)
* Any planned or anticipated surgical treatment for spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in MRI Tractography | Time 0 and after 1 year of treatment
  MRI tractography will be performed at baseline and 1 year post treatment. This imaging modality allows for a detailed picture of the spinal cord motor tracts (the corticospinal tracts). We will measure these tracts (thickness, density, lengths) according to standard tractography protocol and record any change in said measures after treatment.

SECONDARY OUTCOMES:
Change in ASIA motor score over time. | Prior to treatment and after 1 year of treatment
  Assess ASIA standardised motor level of SCI patients

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Stacey, MD, Principal Investigator — McMaster University; Shanker Nesathurai, MD, MPh, Principal Investigator — Hamilton Health Sciences, McMaster University
Locations (1):
- Regional Rehabilitation Centre At Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Pickett GE, Campos-Benitez M, Keller JL, Duggal N. Epidemiology of traumatic spinal cord injury in Canada. Spine (Phila Pa 1976). 2006 Apr 1;31(7):799-805. doi: 10.1097/01.brs.0000207258.80129.03. PMID 16582854
- [Background] Chiu WT, Lin HC, Lam C, Chu SF, Chiang YH, Tsai SH. Review paper: epidemiology of traumatic spinal cord injury: comparisons between developed and developing countries. Asia Pac J Public Health. 2010 Jan;22(1):9-18. doi: 10.1177/1010539509355470. PMID 20032030
- [Background] Hall ED, Wolf DL. A pharmacological analysis of the pathophysiological mechanisms of posttraumatic spinal cord ischemia. J Neurosurg. 1986 Jun;64(6):951-61. doi: 10.3171/jns.1986.64.6.0951. PMID 3084721
- [Background] Hall ED, Braughler JM. Role of lipid peroxidation in post-traumatic spinal cord degeneration: a review. Cent Nerv Syst Trauma. 1986 Fall;3(4):281-94. doi: 10.1089/cns.1986.3.281. PMID 3555850
- [Background] Anderson DK, Demediuk P, Saunders RD, Dugan LL, Means ED, Horrocks LA. Spinal cord injury and protection. Ann Emerg Med. 1985 Aug;14(8):816-21. doi: 10.1016/s0196-0644(85)80064-0. PMID 3927795
- [Background] Robert AA, Zamzami M, Sam AE, Al Jadid M, Al Mubarak S. The efficacy of antioxidants in functional recovery of spinal cord injured rats: an experimental study. Neurol Sci. 2012 Aug;33(4):785-91. doi: 10.1007/s10072-011-0829-4. Epub 2011 Nov 8. PMID 22068217
- [Background] Bastani NE, Kostovski E, Sakhi AK, Karlsen A, Carlsen MH, Hjeltnes N, Blomhoff R, Iversen PO. Reduced antioxidant defense and increased oxidative stress in spinal cord injured patients. Arch Phys Med Rehabil. 2012 Dec;93(12):2223-8.e2. doi: 10.1016/j.apmr.2012.06.021. Epub 2012 Jul 5. PMID 22772083
- [Background] The Incidence and Prevalence of Spinal Cord Injury in Canada: Overview and estimates based on current evidence: Joint publication of Urban Futures and The Rick Hansen Institute. Urban Futures Institute, 2010.